CLINICAL TRIAL: NCT01234701
Title: Agreement Among Expert Radiologists in Diagnosing Primary Liver Tumors by Magnetic Resonance Imaging (MRI) in Non-Cirrhotic Patients - A Double Blind International Multicenter Study
Brief Title: Agreement Among Expert Radiologists in Diagnosing Primary Liver Tumors by Magnetic Resonance Imaging (MRI)
Acronym: MRevaluation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Harvard University (Other); University Hospital, Essen (Other); Auckland City Hospital (Other Government); University Hospital, Strasbourg, France (Other); The Leeds Teaching Hospitals NHS Trust (Other); Imperial College London (Other); University College London Hospitals (Other); St. Louis University (Other)
Responsible Party: Sponsor
Other Study IDs: MRI_Liver_Tumours_Evlauation
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Neoplasms
Keywords: Liver; Neoplasms; Magnetic Resonance Imaging; Surgery; Pathology
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary liver tumors, non-cirrhotic: This single Cohort/Group will include all consecutive patients that received pre-operative Magnetic Resonance Imaging (MRI) and underwent resection for primary liver tumors.
  Interventions: Other: Non-invasive Magnetic Resonance Imaging (MRI); Procedure: Liver resection; Other: Histopathology diagnosis of resected liver specimen

INTERVENTIONS:
Other: Non-invasive Magnetic Resonance Imaging (MRI) — Conventional pre-operative MRI
  Other Names: Magnetic Resonance Imaging
Procedure: Liver resection — Hepatectomy with an intention to cure
  Other Names: Hepatectomy = liver resection by open surgery.
Other: Histopathology diagnosis of resected liver specimen — Histopathology diagnosis by expert pathologist.
  Other Names: Examination under the microscope.

SUMMARY:
The purpose of this multicenter study is to evaluate the agreement among expert radiologists in interpreting magnetic resonance images (MRI) assessing common primary liver tumours in non-cirrhotic patients.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) is currently the method of choice for non-invasive diagnosis of primary liver tumors. However, differentiation of hepatocellular carcinoma (HCC) from adenoma and focal nodular hyperplasia (FNH) remains challenging, particularly in non-cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of Hepatocellular Cancer (HCC), Adenoma and/or Focular nodular hyperplasia (FNH).
* Patients that received a pre-operative Magnetic Resonance Imaging (MRI).
* Patients that underwent liver resection with an intention to cure.
* Patient over 18 years of age

Exclusion Criteria:

* Other histopathological diagnosis such as cysts and hemangiomas.
* Patient age less than 18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Inter-observer agreement among expert radiologists in diagnosing primary liver tumors by Magnetic Resonance Imaging (MRI). | December 2010
  Inter-observer agreement for categorical data will by assessed by the Fliess' kappa (good agreement >0.7).

SECONDARY OUTCOMES:
Agreement of radiologists with the actual diagnosis of primary liver tumors assessed by Magnetic Resonance Imaging (MRI). | December 2010
  The actual diagnosis is defined as the histopathology diagnosis of the resected liver specimen, the current gold standard technique. Such agreement will be assessed by Cohen's Kappa (good agreement >0.7).
Differences in radiologist' certainty of diagnosis (CoD) among different tumor types. | December 2010
  Radiologist' certainty of diagnosis (CoD) will be assessed by a Visual Analogue Scale (VAS 1-10). Potential differences in CoD will be identified by non-parametric multiple comparisons.
Intra-class correlation coefficient among radiologists' Certainty of Diagnosis (CoD) in diagnosis primary liver tumors by Magnetic Resonant Imaging (MRI) | December 2010
  Intra-class correlation coefficient is a descriptive statistic that can be used when quantitative measurements are made on units that are organized into groups. It describes how strongly units in the same group resemble each other.
Investigate the diagnostic efficacy of radiologists' certainty of diagnosis (CoD) in accurately predicting primary liver tumors assessed by Magnetic Resonant Imaging (MRI) | December 2010
  Diagnostic efficacy will be assessed by Receiver Operating Characteristic (ROC) Curves.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, MD, Principal Investigator — University Hospital Zurich, Department of Visceral and Transplant Surgery, Zurich, Switzerland
Locations (10):
- United States (2):
  - Harvard Medical School, Massachusetts General Hospital, and Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Louis University, Liver Center, St Louis, Missouri
- University Hospital Strasbourg, Strasbourg, Cedex, France
- University Hospital Essen, Essen, Germany
- Auckland City Hospital, Auckland, Auckland, New Zealand
- Switzerland (2):
  - University Hospital Zurich, Department of Interventional and Diagnostic Radiology, Zurich, Canton of Zurich
  - University Hospital Zurich, Department of Visceral and Transplant Surgery, Swiss Hepato-Pancreato-Biliary (HPB) Center, Zurich, Canton of Zurich
- United Kingdom (3):
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals NHS Foundation Trust, London
  - Imperial College, Hammersmith Hospital, London

REFERENCES:
- See also: Inter-rater reliability (also called: inter-rater agreement, or concordance) definitions and further information — http://en.wikipedia.org/wiki/Inter-rater_reliability
- See also: Fleiss' kappa information — http://en.wikipedia.org/wiki/Fleiss%27_kappa
- See also: Cohen's kappa information — http://en.wikipedia.org/wiki/Cohen%27s_kappa
- See also: Intraclass correlation information — http://en.wikipedia.org/wiki/Intra-class_correlation_coefficient